CLINICAL TRIAL: NCT01127139
Title: Effectiveness and Patient Self-assessed Compliance of Blood Pressure Treatment With VerapamilSR/ Trandolapril Fixed Combination (Tarka®) in Patients With Essential Hypertension in Routine Clinical Practice
Brief Title: Effectiveness and Patient Self-assessed Compliance of Blood Pressure Treatment With Tarka® Fixed Combination in Patients With Essential Hypertension
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: P12-161
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Results first posted 2012-05-01 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-03

CONDITIONS: Essential Hypertension
Keywords: Essential hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Czech patients with essential hypertension: Czech hypertensive patients (women and men) with systolic blood pressure (SBP) ≥ 140 mmHg or diastolic blood pressure (DBP) ≥ 90 mmHg who can be treated with fixed-combination Tarka®.

SUMMARY:
The fixed combination of verapamil SR/trandolapril (Tarka®) is an effective, well-tolerated therapy for the treatment of essential hypertension in those who require more than one agent to achieve optimal blood pressure (BP) control. The endpoint is compliance with Tarka® treatment by number/percentage of patients continued on fixed combination Tarka therapy after six months. This Post Marketing Observational Study will be conducted in a prospective, single-arm, single-country, multicenter format. The investigational sites will be the cardiologists, the doctors of internal medicine and general practicians. Since this will be a Post Marketing Observational Study, Tarka® will be prescribed in usual manner in accordance with the terms of the local market authorization with regards to dose, population and indication as well as the local guidelines.

DETAILED DESCRIPTION:
Follow-up of patients enables 4 patient visits during this period. For these reasons, the most likely visits are defined as "Inclusion visit" at which treatment with Tarka® is to be initiated, and then "Follow-up visit Week 4-6", "Follow-up visit Month 3 " and "Follow-up visit Month 6", although dates will depend only on the decision of the physician. For these reasons, the most likely visits are defined as "S/V" (Screening Visit), "F1" (Follow-up 1), "F2" (Follow-up 2), "F3" (Follow-up 3). The end point is compliance with Tarka® treatment by number/percentage of patients continued on fixed combination Tarka therapy after six months.

ELIGIBILITY:
Inclusion Criteria:

* Men, women more than 18 years
* Patients with uncontrolled essential hypertension eligible to Tarka treatment according to local label (BP ≥ 140/90 mmHg)
* Patients providing oral informed consent (including consent of their medical data to be used for a Post Marketing Observational Study) and cooperating with physician
* Patients who never received Tarka® in the past
* Patients whom Tarka® will be prescribed according to the labelled indication and dose

Exclusion Criteria:

* Patients contraindicated for treatment of Tarka® according to the local Summary of Product Characteristics (SmPC):
* Hypersensitive to the active substances or to any of the inactive ingredients
* With cardiogenic shock
* With second and third degree atrioventricular block - except in patients with a functioning artificial pacemaker
* With sick sinus syndrome - except in patients with a functioning artificial pacemaker
* With atrial fibrillation/flutter and concomitant Wolff-Parkinson-White syndrome
* With existing history of angioedema associated with administration of an ACE inhibitor
* With severe renal (creatinine clearance < 10 ml/min) or severe liver impairment (cirrhosis with ascites)
* Pregnant women, women of childbearing potential who are unwilling to use contraception
* Lactating women
* Patients who have participated in clinical studies within the last month or who are currently enrolled in clinical studies
* Patients currently treated with other fixed antihypertensive combination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg
Sampling Method: Non-Probability Sample
Enrollment: 3828 (Actual)
Dates: Start 2010-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Hloska, M.D., Study Director — Abbott
Locations (134):
- Czechia (134):
  - Site Reference ID/Investigator# 44896, Babice
  - Site Reference ID/Investigator# 40910, Beroun
  - Site Reference ID/Investigator# 40908, Bílovec
  - Site Reference ID/Investigator# 38816, Blansko
  - Site Reference ID/Investigator# 41189, Brandýs nad Labem
  - Site Ref # / Investigator 40958, Brno
  - Site Reference ID/Investigator# 40821, Brno
  - Site Reference ID/Investigator# 40944, Brno
  - Site Reference ID/Investigator# 41112, Brno
  - Site Reference ID/Investigator# 41187, Brno
  - Site Reference ID/Investigator# 41196, Brno
  - Site Reference ID/Investigator# 44887, Brno
  - Site Reference ID/Investigator# 42083, Brumov
  - Site Reference ID/Investigator# 40967, Bruntál
  - Site Reference ID/Investigator# 40918, Břeclav
  - Site Reference ID/Investigator# 41119, Buštěhrad
  - Site Reference ID/Investigator# 41195, Buštěhrad
  - Site Reference ID/Investigator# 38836, Bystřice nad Pernštejnem
  - Site Reference ID/Investigator# 41190, Bystřice nad Pernštejnem
  - Site Ref # / Investigator 41626, C. Trebova
  - Site Reference ID/Investigator# 42082, Cheb
  - Site Reference ID/Investigator# 41191, České Budějovice
  - Site Ref # / Investigator 38710, České Budějovice
  - Site Reference ID/Investigator# 40948, České Budějovice
  - Site Reference ID/Investigator# 40960, České Budějovice
  - Site Reference ID/Investigator# 40914, České Budějovice
  - Site Reference ID/Investigator# 57305, České Budějovice
  - Site Reference ID/Investigator# 38886, Děčín
  - Site Reference ID/Investigator# 41110, Děčín
  - Site Reference ID/Investigator# 40818, Děčín
  - Site Reference ID/Investigator# 40897, Děčín
  - Site Ref # / Investigator 40902, Děčín
  - Site Reference ID/Investigator# 41117, Hadačka
  - Site Reference ID/Investigator# 40808, Havirov,Ostrava
  - Site Reference ID/Investigator# 41103, Havířov
  - Site Reference ID/Investigator# 40909, Horní Slavkov
  - Site Reference ID/Investigator# 41185, Hradec Králové
  - Site Reference ID/Investigator# 41188, Hradec Králové
  - Site Reference ID/Investigator# 41197, Hranice
  - Site Reference ID/Investigator# 40805, Hranice
  - Site Reference ID/Investigator# 40815, Hranice U Asa
  - Site Reference ID/Investigator# 38736, Jihlava
  - Site Reference ID/Investigator# 38844, Karlovy Vary
  - Site Reference ID/Investigator# 41184, Kdyně
  - Site Reference ID/Investigator# 41113, Kladno
  - Site Ref # / Investigator 44894, Kladno
  - Site Reference ID/Investigator# 40905, Kopřivnice
  - Site Ref # / Investigator 40961, Krnov
  - Site Reference ID/Investigator# 40901, Kunovice
  - Site Reference ID/Investigator# 41192, Kutná Hora
  - Site Reference ID/Investigator# 40811, Litomyšl
  - Site Reference ID/Investigator# 41106, Litvínov
  - Site Reference ID/Investigator# 40904, Louny
  - Site Reference ID/Investigator# 40969, Lovosice
  - Site Reference ID/Investigator# 40953, Malšice
  - Site Reference ID/Investigator# 41204, Mladá Boleslav
  - Site Ref # / Investigator 44882, Mladá Boleslav
  - Site Reference ID/Investigator# 40804, Mnichovo Hradiště
  - Site Ref # / Investigator 41118, Nový Jičín
  - Site Reference ID/Investigator# 40954, Nový Jičín
  - Site Ref # / Investigator 38569, Nymburk
  - Site Reference ID/Investigator# 41114, Olomouc
  - Site Reference ID/Investigator# 40949, Olomouc
  - Site Reference ID/Investigator# 41107, Olomouc
  - Site Ref # / Investigator 40907, Olomouc
  - Site Reference ID/Investigator# 41202, Orlová
  - Site Reference ID/Investigator# 40816, Ostrava
  - Site Reference ID/Investigator# 40951, Ostrava
  - Site Reference ID/Investigator# 40972, Ostrava
  - Site Reference ID/Investigator# 41194, Ostrava
  - Site Reference ID/Investigator# 40968, Ostrava
  - Site Reference ID/Investigator# 40945, Pardubice
  - Site Reference ID/Investigator# 40957, Pardubice
  - Site Reference ID/Investigator# 41201, Pardubice
  - Site Reference ID/Investigator# 41205, Pardubice
  - Site Reference ID/Investigator# 41625, Pardubice
  - Site Reference ID/Investigator# 40956, Pilsen
  - Site Reference ID/Investigator# 40896, Pilsen
  - Site Ref # / Investigator 46282, Pilsen
  - Site Reference ID/Investigator# 40900, Plasy
  - Site Reference ID/Investigator# 41111, Poděbrady
  - Site Ref # / Investigator 40911, Prachatice
  - Site Reference ID/Investigator# 41120, Prague
  - Site Reference ID/Investigator# 41108, Prague
  - Site Reference ID/Investigator# 40822, Prague
  - Site Reference ID/Investigator# 44886, Prague
  - Site Ref # / Investigator 40819, Prague
  - Site Reference ID/Investigator# 40817, Prague
  - Site Reference ID/Investigator# 40812, Prague
  - Site Reference ID/Investigator# 38628, Prague
  - Site Reference ID/Investigator# 44883, Prague
  - Site Reference ID/Investigator# 41193, Prague
  - Site Reference ID/Investigator# 44884, Prague
  - Site Reference ID/Investigator# 40917, Prague
  - Site Reference ID/Investigator# 40913, Prague
  - Site Reference ID/Investigator# 41123, Prague
  - Site Reference ID/Investigator# 41124, Prague
  - Site Reference ID/Investigator# 40903, Prague
  - Site Reference ID/Investigator# 38630, Prague
  - Site Reference ID/Investigator# 40802, Prague
  - Site Reference ID/Investigator# 40823, Prague
  - Site Reference ID/Investigator# 41126, Přelouč
  - Site Reference ID/Investigator# 41198, Přelouč
  - Site Reference ID/Investigator# 40809, Příbram
  - Site Reference ID/Investigator# 40952, Rokycany
  - Site Reference ID/Investigator# 44893, Slaný
  - Site Reference ID/Investigator# 41109, Slatiňany
  - Site Reference ID/Investigator# 40919, Smržovka
  - Site Ref # / Investigator 40807, Stará Paka
  - Site Reference ID/Investigator# 40814, Staré Město
  - Site Reference ID/Investigator# 42085, Staré Město
  - Site Reference ID/Investigator# 41104, Sternberk
  - Site Reference ID/Investigator# 38746, Svitavy
  - Site Reference ID/Investigator# 41121, Tábor
  - Site Ref # / Investigator 40820, Teplice
  - Site Reference ID/Investigator# 40895, Trutnov
  - Site Reference ID/Investigator# 41203, Třanovice
  - Site Reference ID/Investigator# 38739, Třebíč
  - Site Reference ID/Investigator# 40970, Třinec
  - Site Reference ID/Investigator# 40971, Třinec
  - Site Reference ID/Investigator# 41200, Třinec
  - Site Ref # / Investigator 40955, Turnov
  - Site Reference ID/Investigator# 40959, Uherské Hradiště
  - Site Reference ID/Investigator# 41182, Uherské Hradiště
  - Site Reference ID/Investigator# 40906, Ústí nad Labem
  - Site Reference ID/Investigator# 41116, Ústí nad Labem
  - Site Reference ID/Investigator# 40950, Valašské Meziříčí
  - Site Reference ID/Investigator# 40813, Vyškov
  - Site Reference ID/Investigator# 41105, Vyškov
  - Site Ref # / Investigator 41115, Zábřeh
  - Site Reference ID/Investigator# 41186, Zdar
  - Site Reference ID/Investigator# 42084, Zdar
  - Site Reference ID/Investigator# 44895, Zlonice
  - Site Reference ID/Investigator# 40916, Žamberk

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Czech Patients With Essential Hypertension
Started | 3828
Number of Participants Analyzed | 3828
Completed | 3771
Not Completed | 57
Not completed — Adverse Event | 40
Not completed — Incompliance | 12
Not completed — Lack of Efficacy | 4
Not completed — Reason not specified | 1

BASELINE CHARACTERISTICS:
Arm/Group | Czech Patients With Essential Hypertension
Number analyzed (Participants) | 3828
Age, Customized [Number; unit: Participants]
  Age not reported | 3828
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1943
  Male | 1885

OUTCOME MEASURES:

1. Primary Outcome: Compliance With Tarka Treatment, All Participants and by Gender.
Description: Participants were asked how many doses of Tarka they had missed after three months of treatment.
Time Frame: Month 3 Visit
Population: All participants with evaluable case report forms were analyzed.
Measure: Number; unit: participants
Groups:
- Total: Czech hypertensive patients (women and men) with systolic blood pressure (SBP) ≥ 140 mmHg or diastolic blood pressure (DBP) ≥ 90 mmHg treated with fixed-combination Tarka®.
- Female Participants: Female Czech hypertensive patients with systolic blood pressure (SBP) ≥ 140 mmHg or diastolic blood pressure (DBP) ≥ 90 mmHg treated with fixed-combination Tarka®.
- Male Participants: Male Czech hypertensive patients with systolic blood pressure (SBP) ≥ 140 mmHg or diastolic blood pressure (DBP) ≥ 90 mmHg treated with fixed-combination Tarka®.
Arm/Group | Total | Female Participants | Male Participants
Number analyzed (Participants) | 3828 | 1943 | 1885
participants
  Never missed a dose | 2190 | 1141 | 1049
  Missed one dose | 1095 | 548 | 547
  Missed two doses | 446 | 213 | 233
  Missed more than 2 doses | 82 | 41 | 56

2. Secondary Outcome: Change in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: The mean (average) change in participants' systolic blood pressure and diastolic blood pressure from the baseline visit to the Month 6 visit.
Time Frame: Baseline to Month 6 Visit
Population: This analysis included all participants with complete data for the entire study.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Czech Patients With Essential Hypertension
Number analyzed (Participants) | 3783
mmHg
  Change in systolic blood pressure | -28.28 (12.85)
  Change in diastolic blood pressure | -16.39 (9.49)

3. Secondary Outcome: Percentage of Patients Achieving Blood Pressure < 140/90 mmHg
Description: The percentage of patients who had achieved blood pressure less than 140/90 mmHg after three months of treatment.
Time Frame: Month 3 Visit
Population: This analysis included all participants with complete data for the entire study.
Measure: Number; unit: Percentage of participants
Arm/Group | Czech Patients With Essential Hypertension
Number analyzed (Participants) | 3783
Percentage of participants | 44.8

4. Secondary Outcome: Percentage of Patients Achieving Blood Pressure < 140/90 mmHg
Description: The percentage of patients who had achieved blood pressure less than 140/90 mmHg after six months of treatment.
Time Frame: Month 6 Visit
Population: This analysis included all participants with complete data for the entire study.
Measure: Number; unit: Percentage of participants
Arm/Group | Czech Patients With Essential Hypertension
Number analyzed (Participants) | 3783
Percentage of participants | 64.5

5. Secondary Outcome: Number and Type of Antihypertensive Drugs Added to Fixed Combination Tarka to Reach Blood Pressure Goal
Description: The number of participants at the Month 3 visit who were taking other antihypertensive drugs in addition to their Tarka treatment to reach blood a pressure goal of less than 140/90 mmHg. The number of participants taking each type of additional drug is summarized.
Time Frame: Month 3 Visit
Population: This analysis included all participants with complete data for the entire study.
Measure: Number; unit: Participants
Arm/Group | Czech Patients With Essential Hypertension
Number analyzed (Participants) | 3783
Participants
  Central hypotensives | 50
  Angiotensin receptor blockers | 9
  Angiotensin receptor blocker + diuretic | 2
  Angiotensin-converting enzyme (ACE) inhibitors | 6
  Diuretic | 84
  Combined diuretic | 11
  Beta blocker | 8
  Calcium channel blocker | 2

6. Primary Outcome: Compliance With Tarka Treatment, All Participants and by Gender.
Description: Participants were asked how many doses of Tarka they had missed since their previous visit.
Time Frame: Month 6 Visit
Population: All participants with evaluable case report forms were analyzed.
Measure: Number; unit: participants
Arm/Group | Total | Female Participants | Male Participants
Number analyzed (Participants) | 3828 | 1943 | 1885
participants
  Never missed a dose | 2239 | 1181 | 1058
  Missed one dose | 901 | 420 | 481
  Missed two doses | 495 | 253 | 242
  Missed more than 2 doses | 193 | 89 | 104

7. Secondary Outcome: Number and Type of Antihypertensive Drugs Added to Fixed Combination Tarka to Reach Blood Pressure Goal
Description: The number of participants at the Month 6 visit who were taking other antihypertensive drugs in addition to their Tarka treatment to reach a blood pressure goal of less than 140/90 mmHg. The number of participants taking each type of additional drug is summarized.
Time Frame: Month 6 Visit
Population: This analysis included all participants with complete data for the entire study.
Measure: Number; unit: Participants
Arm/Group | Czech Patients With Essential Hypertension
Number analyzed (Participants) | 3783
Participants
  Central hypotensives | 13
  Angiotensin receptor blockers | 4
  Angiotensin receptor blocker + diuretic | 2
  Angiotensin-converting enzyme (ACE) inhibitors | 2
  Diuretic | 23
  Combined diuretic | 1
  Beta blocker | 2

8. Secondary Outcome: Adverse Events Leading to Study Discontinuation
Description: The number of participants who discontinued from the study due to an adverse event and reported event descriptions are summarized.
Time Frame: Baseline to Month 6 Visit
Population: All participants with case report forms were included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Czech Patients With Essential Hypertension
Number analyzed (Participants) | 3828
Participants
  Total discontinued study due to an adverse event | 40
  > Face oedema | 1
  > Nausea | 2
  > Tremor | 1
  > Dyspepsia | 1
  > Feet oedema | 2
  > Allergic reaction | 1
  > Stomach hyperacidity | 1
  > Night cough | 1
  > Constipation | 6
  > Dry cough | 12
  > Hypotension | 3
  > Intolerance | 3
  > Tachycardia | 2
  > Not specified | 1
  > Hypertension | 1
  > Constipation + dry cough + hair loss | 1
  > Rash + palpitation | 1

ADVERSE EVENTS:
Time Frame: Participants were followed for a period of 6 months or until discontinuation of treatment.
Arm/Group | Czech Patients With Essential Hypertension
Serious Adverse Events (participants affected / at risk) | 0/3828
Other Adverse Events (participants affected / at risk) | 0/3828

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.